CLINICAL TRIAL: NCT06301997
Title: Evaluation of Therapeutic Effects of ZAX.1400.P03 a Herbal Compound on Clinical Signs of Skin in Psoriasis Patients
Brief Title: A Herbal Compound for Psoriasis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fasa University of Medical Sciences (Other)
Collaborators: Zarrin Avaye Kowsar Salamat (ZAX company) and HerbmedX (Unknown); Herbmedx Co (Industry)
Responsible Party: Principal Investigator, Akbar Farjadfar, Principle-Investigator, Fasa University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRCT20210218050404N5; IR.FUMS.REC.1400.125 (Other: Fasaums)
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis; Inflammation; Skin Diseases
Keywords: Skin Diseases; Psoriasis; Herbal Medicines; Anti-inflammatory; Natural Products; Inflammation
MeSH Terms: conditions — Psoriasis; Inflammation; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical ZAX.1400.P03 (Experimental): ZAX.1400.P03, applied topically twice daily for 3 weeks after enrolment
  Interventions: Dietary Supplement: ZAX.1400.P03
- Placebo (Placebo Comparator): Placebo, applied topically twice daily for 3 weeks after enrolment
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: ZAX.1400.P03 — ZAX.1400.P03, applied twice daily for 3 weeks after enrolment
  Arms: Topical ZAX.1400.P03
Drug: Placebo — Placebo, applied twice daily for 3 weeks after enrolment
  Arms: Placebo

SUMMARY:
The goal of this interventional clinical trial study is to compare ZAX.1400.P03 and placebo in Psoriasis patients. The main question it aims to answer is:

• Can treatment with ZAX.1400.P03 for 3 weeks improve clinical signs of skin in psoriasis patients? Participants will be divided into two groups of 52 people. One group will use ZAX.1400.P03 topically twice daily for 3 weeks and the other group will use placebo topically twice daily for 3 weeks.

Researchers will compare treatment and placebo groups to see if there is any improvement in the clinical signs of skin caused by psoriasis after treatment with ZAX.1400.P03 for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of the disease by a doctor
* Age range between 18 and 60 years
* Both sexes (male and female)
* Having written informed consent to participate in the study
* Lack of allergy to food and health products
* Only local tissue involvement and no need to take oral medications
* Absence of underlying diseases and immune deficiency
* Absence of pregnancy and breastfeeding
* Absence of blisters and infection caused by the disease

Exclusion Criteria:

* Non-consent of the doctor directly responsible for the patient
* Incidence of drug product allergy
* Occurrence of symptoms of skin, digestive, liver or kidney diseases
* Patient's lack of consent to continue for any reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Dermatology Life Quality Index (DLQI) score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  DLQI score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42

SECONDARY OUTCOMES:
Change From Baseline in Percent Body Surface Area (%BSA) at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Body Surface Area (BSA) is a numerical score used to measure the physician's assessment of the percentage of the participant's total BSA involved with psoriasis. BSA = SQRT ((height (cm) X weight (kg))/3600) BSA is in m2, W is weight in kg, and H is height in cm. Total body Surface Area (BSA) in meters squared %Body Surface Area Affected the "Rule of Nine" was be used
Change From Baseline in erythema score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Erythema score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in Swelling score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Swelling score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in pruritus score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Pruritus score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in flake score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Flake score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in skin dryness score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Skin dryness score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in skin irritation score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Skin irritation score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in pain score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Pain score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in skin scratch score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Skin scratch score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in skin scar score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Skin scar score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in skin thickness score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Skin thickness score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in skin rashes score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Skin rashes score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42

CONTACTS AND LOCATIONS:
Locations (1):
- Fasa university of medical sciences, Fasa, Fars, Iran